CLINICAL TRIAL: NCT00978250
Title: A Multi-Histology Phase II Study of 5-Fluoro-2'-Deoxycytidine With Tetrahydrouridine (FdCyd + THU)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Doroshow, M.D., National Cancer Institute, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090214; 09-C-0214
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Results first posted 2019-12-27 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Head and Neck Neoplasms; Lung Neoplasms; Urinary Bladder Neoplasms; Breast Neoplasms
Keywords: DNA Methylation; Advanced Cancer; Methyltransferase Inhibitor; Epigenetics; Gene Re-Expression; Breast Cancer; Head and Neck Cancer; Lung Cancer; Non-Small Cell Lung Cancer; Bladder Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Urinary Bladder Neoplasms; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — 5-fluoro-2'-deoxycytidine; Tetrahydrouridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 5-Fluro-2'-Deoxycytidine (FdCyd) + Tetrahydrouridine (THU) (Experimental): FdCyd (100 mg/m(2)) + THU (350 mg/m(2)) administered 5 days/week for 2 weeks in 28-day cycles
  Interventions: Drug: 5-Fluoro-2'-Deoxycytidine (FdCyd) + Tetrahydrouridine (THU)

INTERVENTIONS:
Drug: 5-Fluoro-2'-Deoxycytidine (FdCyd) + Tetrahydrouridine (THU) — FdCyd, a fluoropyrimidine nucleoside analog, has a short (10-minute) half-life and is rapidly degraded in vivo by cytidine deaminase. However, co-administration with THU, an inhibitor of cytidine/deoxycytidine deaminase, has been shown to increase the area under the curve (AUC) of the parent compound more than 4-fold. Increased FdCyd exposure allows it to be taken up intracellularly and converted to its triphosphate, which is incorporated into deoxyribonucleic acid (DNA) and inhibits the action of the enzyme DNA methyltransferase (DNMT). Inhibition of DNMT, and in turn DNA methylation, can result in the re-expression of tumor suppressor genes.

SUMMARY:
Background:

* Two experimental drugs, FdCyd (also called 5-fluoro-2'-deoxcytidine), and THU (also called tetrahydrouridine), are undergoing trials to test their effectiveness in treating cancer that has not responded to standard therapies. FdCyd is thought to work by changing how genes work in cancer cells. THU does not have any anticancer effects on its own, but it helps keep the other drug, FdCyd, from being broken down by the body.
* These drugs are being tested in several separate clinical trials.

Objectives:

* To determine if FdCyd and THU can work together to control tumor growth.
* To evaluate the safety and tolerability of FdCyd and THU when given together.

Eligibility:

- Individuals 18 years of age and older who have advanced non-small cell lung cancer, breast cancer, bladder cancer, or head and neck cancer that has progressed after receiving standard treatment or for which no effective therapy exists.

Design:

* The drugs are given over 28-day periods called cycles. FdCyd and THU are given through a vein for about 3 hours each day on days 1, 5 and 8, 12 of each cycle.
* Clinical Center visits: FdCyd and THU will be given through a vein on days 1, 5 and 8, 12 of each cycle. During the Clinical Center visits, researchers will perform study tests and procedures to see how the study drugs are affecting the body.
* Patients will undergo a number of tests and procedures during the treatment cycle, including physical examinations, blood and urine samples for standard tests, imaging studies (ultrasound, magnetic resonance imaging (MRI) or computed tomography (CT) scans) to evaluate tumor growth, and blood and urine samples to evaluate the amount of FdCyd and THU in the body and the body's response to the drugs.
* Patients may continue to receive FdCyd and THU if their cancer does not grow, if they do not have too many side effects, and if they are willing to do so.

DETAILED DESCRIPTION:
Background:

5-Fluoro-2'-deoxycytidine (FdCyd), a fluoropyrimidine nucleoside analog, has a short (10-minute) half-life and is rapidly degraded in vivo by cytidine deaminase. However, coadministration with tetrahydrouridine (THU), an inhibitor of cytidine/deoxycytidine deaminase, has been shown to increase the area under the curve (AUC) of the parent compound more than 4-fold. Increased FdCyd exposure allows it to be taken up intracellularly and converted to its triphosphate, which is incorporated into deoxyribonucleic acid (DNA) and inhibits the action of the enzyme DNA methyltransferase (DNMT). Inhibition of DNMT, and in turn DNA methylation, can result in the re-expression of tumor suppressor genes.

Primary objective:

-Determine progression-free survival (PFS) and/or the response rate (Complete Response (CR) + Partial Response (PR)) of FdCyd administered 5 days per week for 2 weeks, in 28-day cycles, by intravenous infusion over 3 hours along with THU in patients with breast cancer, head and neck cancer, non-small cell lung cancer (NSCLC), and urothelial transitional cell carcinoma.

Exploratory objectives:

* Evaluate whether treatment with FdCyd and THU alters DNA methylation patterns in tumor biopsy samples before and during treatment by long interspersed nuclear element-1 (LINE-1) analysis.
* Evaluate the safety and tolerability of FdCyd (100 mg/m(2)) + THU (350 mg/m(2)) administered 5 days per week for 2 weeks, in 28-day cycles, by intravenous infusion over 3 hours.
* Measure changes in the number of circulating tumor cells (CTCs) following treatment with FdCyd plus THU.

Eligibility:

-Patients with histologically documented non-small cell lung cancer, head and neck cancer, urothelial transitional cell carcinoma, and breast carcinoma.

Design:

* This is a multicenter trial with National Cancer Institute (NCI) as the coordinating center and the California Cancer Consortium and University of Pittsburgh Medical Center (UPMC) as participating sites.
* FdCyd will be administered as an intravenous (IV) infusion over 3 hours with 20% of the daily dose of THU administered as an IV push and the remaining 80% co-administered with FdCyd by 3-hour infusion daily for 5 consecutive days of treatment per week for 2 consecutive weeks, followed by 2 weeks of no treatment, in a 28-day cycle.
* Blood and optional tumor biopsies for pharmacodynamic and pharmacokinetic studies will be obtained.
* The study will accrue a maximum of 165 patients including all centers.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically documented metastatic or unresectable non-small cell lung cancer, head and neck cancer, urothelial transitional cell carcinoma, or breast cancer whose disease has progressed after at least one line of standard therapy.
* Patients with solid tumors (non-small cell lung cancer, head and neck cancer, urothelial transitional cell carcinoma, and breast cancer) must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as greater than or equal to 20 mm with conventional techniques or as greater than or equal 10 mm with spiral computed tomography (CT) scan. Patients with the above tumor types whose disease is limited to the skin are eligible at the discretion of the principal investigator (PI) and must have a physical exam with documentation of skin lesion(s) by color photography, including a ruler to estimate the size of the lesion(s).
* Diagnosis of malignancy must be confirmed by the department of pathology at the institution where the patient is enrolled prior to patient enrollment.
* Any prior therapy must have been completed greater than or equal to 4 weeks prior to enrollment on protocol and the participant must have recovered to eligibility levels from prior toxicity. Patients should be at least six weeks out from nitrosoureas and mitomycin C. Prior radiation should have been completed greater than or equal to 4 weeks prior to study enrollment and all associated toxicities resolved to eligibility levels. Patients must be greater than or equal to 2 weeks since any investigational agent administered as part of a Phase 0 study (also referred to as an "early Phase I study" or "pre-Phase I study" where a sub-therapeutic dose of drug is administered) at the PI's discretion, and should have recovered to eligibility levels from any toxicities.
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of 5-Fluoro-2'-Deoxycytidine (FdCyd) and Tetrahydrouridine (THU) in patients less than 18 years of age, children are excluded from this study, but may be eligible for future pediatric Phase I combination trials.
* Karnofsky performance status greater than or equal to 60%.
* Life expectancy of greater than 3 months.
* Patients must have normal organ and marrow function as defined below:

  * absolute neutrophil count greater than or equal to 1,500/mcL
  * platelets greater than or equal to 100,000/mcL
  * total bilirubin less than 1.5 times institutional upper limit of normal
  * Aspartate transaminase (AST)(Serum glutamic-oxaloacetic transaminase (SGOT))/Alanine transaminase (ALT)(Serum glutamic pyruvic transaminase (SGPT)) less than or equal to 3 times institutional upper limit of normal; less than or equal to 5 times upper limit of normal (ULN) for patients with liver metastases

creatinine less than 1.5 times institutional upper limit of normal

OR

creatinine clearance greater than or equal to 60 mL/min for patients with creatinine levels above 1.5 times institutional upper limit of normal.

* Because FdCyd has been shown to be teratogenic in animals, pregnant women will be excluded from this trial. Nursing women are also excluded, as there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with FdCyd. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation, and for 3 months after completion of study. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she or her partner should inform the treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.
* Patients should not be receiving any other investigational agents.

EXCLUSION CRITERIA:

* Patients with clinically significant illnesses which would compromise participation in the study, including, but not limited to: active or uncontrolled infection, immune deficiencies or confirmed diagnosis of human immunodeficiency virus (HIV) infection, active infection with Hepatitis B or Hepatitis C, uncontrolled diabetes, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmia; or psychiatric illness/social situations that would limit compliance with study requirements.
* History of allergic reactions attributed to fluoropyrimidines (e.g., capecitabine, fluorouracil, fluorodeoxyuridine) or tetrahydrouridine.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2009-08-20 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James H Doroshow, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (4):
- United States (4):
  - University of California, Davis, Davis, California
  - City of Hope National Medical Center, Duarte, California
  - City of Hope Medical Group, South Pasadena, California
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lapeyre JN, Becker FF. 5-Methylcytosine content of nuclear DNA during chemical hepatocarcinogenesis and in carcinomas which result. Biochem Biophys Res Commun. 1979 Apr 13;87(3):698-705. doi: 10.1016/0006-291x(79)92015-1. No abstract available. PMID 454420
- [Background] Herman JG, Baylin SB. Gene silencing in cancer in association with promoter hypermethylation. N Engl J Med. 2003 Nov 20;349(21):2042-54. doi: 10.1056/NEJMra023075. No abstract available. PMID 14627790
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Murray T, Thun MJ. Cancer statistics, 2008. CA Cancer J Clin. 2008 Mar-Apr;58(2):71-96. doi: 10.3322/CA.2007.0010. Epub 2008 Feb 20. PMID 18287387
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-C-0214.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-Small Cell Lung Cancer Stratum; Breast Cancer Stratum; Bladder Cancer Stratum; Head and Neck Cancer Stratum: FdCyd (100 mg/m(2)) + THU (350 mg/m(2)) administered 5 days/week for 2 weeks in 28-day cycles.
Period: Overall Study
Arm/Group | Non-Small Cell Lung Cancer Stratum | Breast Cancer Stratum | Bladder Cancer Stratum | Head and Neck Cancer Stratum
Started | 25 | 30 | 18 | 22
Completed | 25 | 29 | 18 | 21
Not Completed | 0 | 1 | 0 | 1
Not completed — Late determination of ineligibility | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Non-Small Cell Lung Cancer Stratum; Breast Cancer Stratum; Bladder Cancer Stratum; Head and Neck Cancer Stratum: FdCyd (100 mg/m(2)) + THU (350 mg/m(2)) administered 5 days/week for 2 weeks in 28-day cycles
  5-Fluoro-2'-Deoxycytidine (FdCyd) + Tetrahydrouridine (THU): FdCyd, a fluoropyrimidine nucleoside analog, has a short (10-minute) half-life and is rapidly degraded in vivo by cytidine deaminase. However, co-administration with THU, an inhibitor of cytidine/deoxycytidine deaminase, has been shown to increase the area under the curve (AUC) of the parent compound more than 4-fold. Increased FdCyd exposure allows it to be taken up intracellularly and converted to its triphosphate, which is incorporated into deoxyribonucleic acid (DNA) and inhibits the action of the enzyme DNA methyltransferase (DNMT). Inhibition of DNMT, and in turn DNA methylation,can result in the re-expression of tumor suppressor genes.
- Total: Total of all reporting groups
Arm/Group | Non-Small Cell Lung Cancer Stratum | Breast Cancer Stratum | Bladder Cancer Stratum | Head and Neck Cancer Stratum | Total
Number analyzed (Participants) | 25 | 30 | 18 | 22 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 24 | 4 | 16 | 61
  >=65 years | 8 | 6 | 14 | 6 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.92 (9.95) | 56.04 (10.07) | 67.77 (8.93) | 55.17 (11.70) | 59.08 (11.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 30 | 3 | 3 | 45
  Male | 16 | 0 | 15 | 19 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 10 | 1 | 2 | 13
  Not Hispanic or Latino | 25 | 20 | 17 | 20 | 82
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 3 | 3 | 3 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 0 | 2 | 9
  White | 16 | 22 | 15 | 17 | 70
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 30 | 18 | 22 | 95

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the time interval from start of treatment to documented evidence of disease progression. Disease progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) and is at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum of the LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: until subject progressed or went off study for other reasons (up to approximately 1 year)
Population: All 93 patients eligible for the study were assessed for PFS, including patients with advanced non-small cell lung cancer, breast cancer, bladder cancer, or head and neck cancer. Two patients were determined ineligible for the study and never received study drug.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Non-Small Cell Cancer Stratum; Breast Cancer Stratum; Bladder Cancer Stratum; Heand and Neck Cancer Stratum: FdCyd (100 mg/m(2)) + THU (350 mg/m(2)) administered 5 days/week for 2 weeks in 28-day cycles
  5-Fluoro-2'-Deoxycytidine (FdCyd) + Tetrahydrouridine (THU): FdCyd, a fluoropyrimidine nucleoside analog, has a short (10-minute) half-life and is rapidly degraded in vivo by cytidine deaminase. However, co-administration with THU, an inhibitor of cytidine/deoxycytidine deaminase, has been shown to increase the area under the curve (AUC) of the parent compound more than 4-fold. Increased FdCyd exposure allows it to be taken up intracellularly and converted to its triphosphate, which is incorporated into deoxyribonucleic acid (DNA) and inhibits the action of the enzyme DNA methyltransferase (DNMT). Inhibition of daunomycin DNMT, and in turn DNA methylation, can result in the re-expression of tumor suppressor genes.
Arm/Group | Non-Small Cell Cancer Stratum | Breast Cancer Stratum | Bladder Cancer Stratum | Heand and Neck Cancer Stratum
Number analyzed (Participants) | 25 | 29 | 18 | 21
months | 2.3 [1.6 to 3.9] | 3.7 [1.8 to 5.3] | 3.6 [1.7 to 8.0] | 1.7 [1.7 to 4.5]

2. Primary Outcome: Percentage of Participants With (Complete Response (CR) + Partial Response (PR)) to 5-Fluro-2'-Deoxycytidine (FdCyd)
Description: Response was measured using the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response is disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum of the LD.
Time Frame: until subject progressed or went off study for other reasons (up to approximately 1 year)
Population: All 93 patients eligible for the study were assessed for complete response (CR) or partial response (PR), including patients with advanced non-small cell lung cancer, breast cancer, bladder cancer, or head and neck cancer. Two patients were determined ineligible for the study and never received study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Non-Small Cell Cancer Stratum; Breast Cancer Stratum; Bladder Cancer Stratum; Head and Neck Cancer Stratum: FdCyd (100 mg/m(2)) + THU (350 mg/m(2)) administered 5 days/week for 2 weeks in 28-day cycles
  5-Fluoro-2'-Deoxycytidine (FdCyd) + Tetrahydrouridine (THU): FdCyd, a fluoropyrimidine nucleoside analog, has a short (10-minute) half-life and is rapidly degraded in vivo by cytidine deaminase. However, co-administration with THU, an inhibitor of cytidine/deoxycytidine deaminase, has been shown to increase the area under the curve (AUC) of the parent compound more than 4-fold. Increased FdCyd exposure allows it to be taken up intracellularly and converted to its triphosphate, which is incorporated into deoxyribonucleic acid (DNA) and inhibits the action of the enzyme DNA methyltransferase (DNMT). Inhibition of DNMT, and in turn DNA methylation, can result in the re-expression of tumor suppressor genes.
Arm/Group | Non-Small Cell Cancer Stratum | Breast Cancer Stratum | Bladder Cancer Stratum | Head and Neck Cancer Stratum
Number analyzed (Participants) | 25 | 29 | 18 | 21
percentage of participants | 0.0 [0.0 to 13.7] | 6.9 [0.8 to 22.8] | 5.6 [0.1 to 27.3] | 0.0 [0.0 to 16.1]

3. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0).
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 109 months and 16 days.
Population: Two patients were determined ineligible for the study and never received study drug. Adverse Events are not being reported by stratum because this was not specified in the protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | 5-Fluro-2'-Deoxycytidine (FdCyd) + Tetrahydrouridine (THU)
Number analyzed (Participants) | 93
Participants | 91

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 109 months and 16 days. Two patients were determined ineligible for the study and never received study drug.
Description: Adverse Events are not being reported by stratum because this was not specified in the protocol.
Arm/Group | 5-Fluro-2'-Deoxycytidine (FdCyd) + Tetrahydrouridine (THU)
All-Cause Mortality (participants affected / at risk) | 8/93
Serious Adverse Events (participants affected / at risk) | 38/93
Other Adverse Events (participants affected / at risk) | 91/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5-Fluro-2'-Deoxycytidine (FdCyd) + Tetrahydrouridine (THU) (N=93)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (7)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 4 (5)
Anorexia (Metabolism and nutrition disorders) | 2 (3)
Anxiety (Psychiatric disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Death NOS (General disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 4 (6)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 5 (5)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 3 (3)
Gastrointestinal disorders - Other, Diverticulitis (Gastrointestinal disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (4)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Infections and infestations - Other, port infection (right) (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 3 (3)
Lymphocyte count decreased (Investigations) | 6 (6)
Mucosal infection (Infections and infestations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Multi-organ failure (General disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) — Death due to disease progression.
Nervous system disorders - Other, Bilateral lower extremity weakness/paraplegia (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (6)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Platelet count decreased (Investigations) | 3 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Retinopathy (Eye disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (5)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 5 (6)
Gastrointestinal disorders - Other, Pyloric ulcer (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, Partial small bowel obstruction (Gastrointestinal disorders) | 1 (1)
Infections and infestations - Other, Clostridium difficile (Infections and infestations) | 1 (1)
Infections and infestations - Other, Viral syndrome (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5-Fluro-2'-Deoxycytidine (FdCyd) + Tetrahydrouridine (THU) (N=93)
Abdominal distension (Gastrointestinal disorders) | 3 (6)
Abdominal infection (Infections and infestations) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 20 (34)
Activated partial thromboplastin time prolonged (Investigations) | 12 (13)
Agitation (Psychiatric disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 34 (83)
Alkaline phosphatase increased (Investigations) | 26 (49)
Allergic reaction (Immune system disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 62 (196)
Anorexia (Metabolism and nutrition disorders) | 37 (65)
Anxiety (Psychiatric disorders) | 6 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Ascites (Gastrointestinal disorders) | 1 (4)
Aspartate aminotransferase increased (Investigations) | 36 (78)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (20)
Bloating (Gastrointestinal disorders) | 5 (5)
Blood and lymphatic system disorders - Other, Adenopathy: supraclavicular node (Blood and lymphatic system disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 8 (12)
Blurred vision (Eye disorders) | 2 (2)
Body odor (Skin and subcutaneous tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Bruising (Injury, poisoning and procedural complications) | 2 (3)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
CPK increased (Investigations) | 4 (10)
Cardiac troponin I increased (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (6)
Chills (General disorders) | 13 (18)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 3 (6)
Conjunctivitis infective (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 35 (47)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (30)
Creatinine increased (Investigations) | 14 (29)
Dehydration (Metabolism and nutrition disorders) | 12 (17)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (4)
Diarrhea (Gastrointestinal disorders) | 36 (81)
Dizziness (Nervous system disorders) | 12 (13)
Dry eye (Eye disorders) | 2 (4)
Dry mouth (Gastrointestinal disorders) | 8 (10)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (11)
Dysarthria (Nervous system disorders) | 1 (1)
Dysesthesia (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 9 (10)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Nervous system disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 24 (37)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 23 (25)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 2 (3)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Eye disorders - Other, Non-visibility spots, eye stain (Eye disorders) | 1 (1)
Eye disorders - Other, Visual changes (Eye disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (8)
Fatigue (General disorders) | 62 (188)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 23 (53)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Flatulence (Gastrointestinal disorders) | 2 (2)
Flu like symptoms (General disorders) | 6 (7)
Gait disturbance (General disorders) | 4 (4)
Gastritis (Gastrointestinal disorders) | 2 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Gastrointestinal disorders - Other, "pin point" ulcer on tongue (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6 (6)
Genital edema (Reproductive system and breast disorders) | 1 (1)
Gum infection (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 13 (16)
Hematuria (Renal and urinary disorders) | 3 (4)
Hemoglobin increased (Investigations) | 2 (4)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hepatobiliary disorders - Other, Cirrhosis (Hepatobiliary disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 17 (31)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (27)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 8 (20)
Hypermagnesemia (Metabolism and nutrition disorders) | 9 (12)
Hypernatremia (Metabolism and nutrition disorders) | 4 (5)
Hypertension (Vascular disorders) | 29 (175)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 61 (174)
Hypocalcemia (Metabolism and nutrition disorders) | 20 (45)
Hypoglycemia (Metabolism and nutrition disorders) | 8 (8)
Hypokalemia (Metabolism and nutrition disorders) | 23 (47)
Hypomagnesemia (Metabolism and nutrition disorders) | 24 (58)
Hyponatremia (Metabolism and nutrition disorders) | 49 (115)
Hypophosphatemia (Metabolism and nutrition disorders) | 26 (49)
Hypotension (Vascular disorders) | 13 (21)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
INR increased (Investigations) | 4 (6)
Infections and infestations - Other, C. difficile infection (Infections and infestations) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 2 (2)
Injection site reaction (General disorders) | 5 (5)
Insomnia (Psychiatric disorders) | 8 (8)
Investigations - Other, Bicarbonate, serum-low (Investigations) | 4 (5)
Lethargy (Nervous system disorders) | 1 (1)
Lip infection (Infections and infestations) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Lymphedema (Vascular disorders) | 2 (2)
Lymphocyte count decreased (Investigations) | 60 (265)
Malaise (General disorders) | 2 (2)
Memory impairment (Nervous system disorders) | 2 (6)
Mucosal infection (Infections and infestations) | 2 (3)
Mucositis oral (Gastrointestinal disorders) | 9 (13)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal and connective tissue disorder - Other, locking of fingers-middle and ring (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Nail infection (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 57 (107)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Nervous system disorders) | 1 (1) — Drainage/bleeding @ chest mass.
Nervous system disorders - Other, saddle anesthesia (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 28 (76)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 15 (25)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (18)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 (5)
Paresthesia (Nervous system disorders) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Penile infection (Infections and infestations) | 1 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (14)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Platelet count decreased (Investigations) | 37 (91)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Proteinuria (Renal and urinary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (11)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 (12)
Renal and urinary disorders - Other, renal insufficiency (Renal and urinary disorders) | 1 (1)
Renal calculi (Renal and urinary disorders) | 1 (1)
Reproductive system and breast disorders - Other, Orchitis (Reproductive system and breast disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Scleral disorder (Eye disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (3)
Sinus tachycardia (Cardiac disorders) | 11 (34)
Sinusitis (Infections and infestations) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Blisters (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Skin and subcutaneous tissue disorder
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Infections and infestations) | 2 (3)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2)
Somnolence (Nervous system disorders) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 1 (1)
Surgical and medical procedures - Other, hip surgery (Surgical and medical procedures) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 3 (4)
Tinnitus (Ear and labyrinth disorders) | 2 (2)
Tremor (Nervous system disorders) | 2 (2)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Urinary frequency (Renal and urinary disorders) | 3 (4)
Urinary retention (Renal and urinary disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 7 (10)
Urinary tract pain (Renal and urinary disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2)
Vaginal infection (Infections and infestations) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 27 (38)
Watering eyes (Eye disorders) | 3 (4)
Weight gain (Investigations) | 1 (2)
Weight loss (Investigations) | 26 (41)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
White blood cell decreased (Investigations) | 49 (181)
Wound infection (Infections and infestations) | 1 (1)
Gastrointestinal disorders - Other, Blood in stool (Gastrointestinal disorders) | 1 (1)
Infections and infestations - Other, Herpes (Infections and infestations) | 1 (1)
Infections and infestations - Other, Cryptosporidium (Infections and infestations) | 1 (1)
Infections and infestations - Other, C. difficile colitis (Infections and infestations) | 1 (1)
Infections and infestations - Other, catheter related (Infections and infestations) | 1 (1)
Infections and infestations - Other, Infection with unknown ANC: Blood (Infections and infestations) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, Swelling - right arm (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, chest tightness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, hip pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Complex multiseptated cysts - left testicle
Nervous system disorders - Other, disk replacement (Nervous system disorders) | 1 (1)
Renal and urinary disorders - Other, urinary output decreased (Renal and urinary disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, nasal drainage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, facial erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, scleroderma @ hands and feet (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, nail changes (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, discoloration of leg (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, rash (Skin and subcutaneous tissue disorders) | 1 (1)
Infections and infestations - Other, Sinusitis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/50/NCT00978250/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/50/NCT00978250/ICF_001.pdf